CLINICAL TRIAL: NCT00606671
Title: Insulin Resistance in Polycystic Ovary Syndrome (PCOS)
Brief Title: Metabolic Disturbances in Polycystic Ovary Syndrome (PCOS)
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Diabetesforeningen (Other); Danish Hospital foundation for medical research. region Copenhagen, The Faroe Islands and Greenland. (Unknown); Aage Bangs Fond (Other)
Responsible Party: Lisbeth Nilas, Dpt. of Obstetrics and Gynaecology, Copenhagen University Hospital, Hvidovre
Other Study IDs: PCOS
Record Dates: First submitted 2008-01-17; First posted 2008-02-04 (Estimated); Last update posted 2008-02-04 (Estimated); Status verified 2008-01

CONDITIONS: Polycystic Ovary Syndrome
Keywords: polycystic ovary syndrome (PCOS)
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fat and muscle biopsies
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (8):
- 1: lean control women without PCOS
- 2: lean women with PCOS
- 3: Obese control women without PCOS
- 4: Obese women with PCOS
- 1xx - 04 LC: lean control women
- 1xx-04 LP: lean women with PCOS
- 1xx-04 OC: obese control women
- 1xx-04 OP: obese women with PCOS

SUMMARY:
The scope of the study was to investigate different metabolic aspects that may lead to or are a consequence of insulin resistance in premenopausal women with polycystic ovary syndrome (PCOS). We use gold standard methods for evaluation of insulin resistance. We take muscle and fat biopsies for investigation of gene expression of different cytokines associated with insulin resistance. We investigate the incretin hormones GIP and GLP-1. These two hormones play a central role in glycemic control, and diabetic subjects are known to have alterations in their incretin hormones. The incretin hormones have not previously been investigated in women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women that meet the Rotterdam criteria for PCOS (BMI < 40)
* Age and BMI matched control women that do not have any signs or symptoms of PCOS

Exclusion Criteria:

* BMI > 40. mani fest diabetes or other known diseases

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: lean and obese women with and without PCOS
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2004-02; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
insulin resistance | 2004-2006

SECONDARY OUTCOMES:
gene expression of cytokines in fatty tissue | 2004-2006

CONTACTS AND LOCATIONS:
Overall Officials: Pernille Fog Svendsen, MD, Principal Investigator — Dpt. of Obstetrics and Gynaecology, Copenhagen University Hospital, Hvidovre
Locations (1):
- Dpt. of Obstetrics and Gynaecology, Copenhagen University Hospital, Hvidovre, Hvidovre, Denmark